CLINICAL TRIAL: NCT01703533
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Escalation Study of NNZ-2566 in Rett Syndrome
Brief Title: A Safety Study of NNZ-2566 in Patients With Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Collaborators: Baylor College of Medicine (Other); International Rett Syndrome Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-RETT-001
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Rett Syndrome
Keywords: Autism; Rett's Syndrome; Rett Disorder; Rett's Disorder; Ataxia
MeSH Terms: conditions — Rett Syndrome; Autistic Disorder; Ataxia | interventions — trofinetide; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNZ-2566 (Experimental): Glycyl-L-2-Methylpropyl-L-Glutamic Acid
  Interventions: Drug: NNZ-2566
- Placebo (strawberry flavored solution) (Placebo Comparator): Strawberry flavored solution and Water for Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylpropyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder (2g in 50mL vials) for reconstitution with strawberry flavored solution 0.5% v/v in Water for Injection.
  Arms: NNZ-2566
Drug: Placebo — Strawberry flavored solution and Water for Injection
  Other Names: Strawberry flavored solution 0.5% v/v in Water for Injection
  Arms: Placebo (strawberry flavored solution)

SUMMARY:
The purpose of this study is to determine whether NNZ-2566 is safe and well tolerated in the treatment of Rett Syndrome in adolescent and adult females.

DETAILED DESCRIPTION:
Rett Syndrome is a developmental disorder primarily if not exclusively affecting females. The disorder is characterized by apparent normal development in early infancy (6-18 months), followed by a period of regression with onset of systemic and neurological signs. The CNS symptoms of Rett Syndrome include learning disability, autism and epilepsy and these can be severe and highly debilitating. Affected individuals also show signs of autonomic dysfunction, reflected in cardiovascular and respiratory abnormalities. There is no currently effective treatment for Rett Syndrome.

This study will investigate the safety and tolerability of treatment with oral administration of NNZ-2566 at 35 mg/kg or 70 mg/kg BID in adolescent or adult females with Rett Syndrome. The study also will also investigate measures of efficacy during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rett Syndrome with proven mutation of the MeCP2 gene
* Age 16 to 45 years
* Severity rating of between 10 and 36 (Rett Syndrome Natural History/Clinical Severity Scale)
* Concomitant medications must be stable for >4 weeks prior to enrollment. The following concomitant medications are permitted: anticonvulsants which do not have liver inducing effects; beta-blockers; medications for the treatment of gastroesophageal reflux disease (GERD); medications for the treatment of chronic respiratory conditions such as asthma; medications for the treatment of anxiety, of depression and of psychosis, hormonal contraceptives. Melatonin for difficulties with sleep onset.
* Ability to swallow study medication provided as a liquid solution, or via gastrostomy tube

Exclusion Criteria:

* No detectable abnormality of the EEG during screening period
* Actively undergoing regression
* QTcF exclusions (any of the following): baseline/screening QT/QTcF interval of 450 msec; history of risk factors for torsade de pointes (e.g. heart failure, hypokalemia (serum potassium at screening < 3.0 mmol/L) or family history of long QT syndrome; QT/QTcF prolongation previously or currently controlled with medication
* Current treatment with insulin
* Hgb A1C values outside the normal reference range at screening
* Current or past treatment with IGF-1
* Current or past treatment with growth hormone
* Current treatment with N-methyl-D-aspartate (NMDA) antagonists
* Current or planned use of non-medication based interventional therapy during the period of the study (defined as 4-6 week screening period followed by 4 week dosing and 2 week follow-up period)
* Current clinically significant cardiovascular, renal, hepatic or respiratory disease
* Gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the the study medication
* History of, or current cerebrovascular disease or brain trauma
* History of, or current significant endocrine disorder e.g. hypo or hyperthyroidism or diabetes mellitus
* History of, or current malignancy
* Clinically significant abnormalities in safety laboratory tests, vital signs or ECG, as measured at screening or baseline
* Confirmed pregnancy
* Significant hearing and/or visual impairment that may affect ability to complete the test procedures
* Enrollment in another clinical trial within the previous 30 days
* Previously randomized in this clinical trial
* Allergy to strawberries

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adverse events | Through to Day 40
  Incidence of adverse events (AE), including Serious adverse events (SAE), will be evaluated between the two NNZ-2566 doses and placebo. SAEs will be examined from randomization through to Day 40. AEs will be examined from dosing through to Day 40.

SECONDARY OUTCOMES:
Change in EEG activity | Baseline through to Day 40
  Absolute change in the number of spikes in the EEG per hour during the awake state will be calculated for each subject between baseline (pre-treatment), during treatment (Days 1 thru 4, 14 and 26) and after treatment (Day 40).
  Absolute change in the power of frequency bands in the EEG over an hour in the awake state as determined by the Fast Fourier method will be calculated for each subject between baseline (pre-treatment), during treatment (Days 1 thru 4, 14 and 26) and after treatment (Day 40).
  Changes in the frequency of the characteristic repetitive stereotypic hand movements during wakefulness will be calculated for each subject between baseline (pre-treatment), during treatment (Days 1 thru 4, 14 and 26) and after treatment (Day 40).
Behavior | Baseline through to Day 40
  The following measures will be assessed at baseline and Day 26 and the changes compared between active and placebo groups:
  Symptom severity according to the Rett Syndrome Natural History Motor Behavior Assessment (MBA), Clinical Severity Scale (CSS), Aberrant Behavior Checklist (ABC), Vineland Adaptive Behavior Scale (VABS), and Clinical Global Impression of Severity (CGI-S).
  The following assessments will be undertaken at the additional time points specified: CGI-S (screening, baseline, Days 5, 14, 26, and 40), CGI-I (Days 5, 14, 26, and 40), MBA (Baseline, Days 26 and 40), CSS (screening, baseline, Days 26, and 40).
Physiological changes | Baseline through to Day 40
  Changes in autonomic function, i.e. respiratory rhythm, hyperventilation, apneas, oxygen desaturation, and heart rate variation will be calculated between baseline (pre-treatment), during treatment (Days 1 thru 4, 14 and 26) and after treatment (Day 40).
Global and Functional outcome Measures | Baseline through to Day 40
  Global outcome as measured by the change in scores on the Rett Syndrome Clinical Severity Score (CSS), The Rett Syndrome Motor-Behavior Assessment Scale (MBA), and the Clinical Global Impression - Severity and Improvement scales (CGI-S and -I) from baseline, during treatment, and post treatment.
  Changes in caregiver assessment of the top three causes for concern as assessed via a Visual Analogue Scale (VAS) will be evaluated for each subject between baseline (pre-treatment), during treatment (Day 26) and after treatment (Day 40).
  Changes in the Aberrant Behavior Checklist (ABC) and Vineland Adaptive Behavior Scales (VABS) will be calculated for each subject between baseline (pre-treatment), and during treatment (Day 26).

OTHER OUTCOMES:
Pharmacokinetics | Baseline through to Day 40
  The following pharmacokinetic measures will be calculated from NNZ-2566 concentrations in whole blood: Tmax, Cmax (peak), Cmin (trough), CAV at steady state, T1/2 and AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Glaze, M.D., Principal Investigator — Baylor College of Medicine; Jeffrey L Neul, M.D., Ph.D., Principal Investigator — Baylor College of Medicine; Alan Percy, MD, Principal Investigator — University of Alabama at Birmingham; Timothy Feyma, MD, Principal Investigator — Gillette Children's Specialty Healthcare; Arthur Beisang, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Baylor School of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Darwish M, Passarell J, Youakim JM, Bradley H, Bishop KM. Exposure-Response Efficacy Modeling to Support Trofinetide Dosing in Individuals with Rett Syndrome. Adv Ther. 2024 Apr;41(4):1462-1480. doi: 10.1007/s12325-024-02796-y. Epub 2024 Feb 16. PMID 38363467
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385